CLINICAL TRIAL: NCT06221592
Title: Differences and Wearing Safety and Comfort of New Defocus Incorporated Multiple Segments Spectacle Lenses in Myopia Prevention and Control
Brief Title: Differences and Wearing Safety and Comfort of New Defocus Incorporated Multiple Segments Spectacle Lenses
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: Shanghai Eye Disease Prevention and Treatment Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: QX-2023-A-03
Record Dates: First submitted 2023-12-17; First posted 2024-01-24 (Actual); Last update posted 2024-10-01 (Actual); Status verified 2024-01

CONDITIONS: Myopia, Progressive
MeSH Terms: conditions — Myopia, Degenerative

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (4):
- Full axis multi-point defocus spectacle lenses (Experimental)
  Interventions: Device: defocus spectacle lenses
- Innovative micro defocus spectacle lenses (Experimental)
  Interventions: Device: defocus spectacle lenses
- Circular multi-point optical micro transparent defocus spectacle lenses (Experimental)
  Interventions: Device: defocus spectacle lenses
- High non spherical micro transparent defocus spectacle lenses (Placebo Comparator)
  Interventions: Device: defocus spectacle lenses

INTERVENTIONS:
Device: defocus spectacle lenses — To evaluate the differences in controlling the progression of myopia in adolescents and the safety and comfort of wearing different types of defocus incorporated multiple segments spectacle lenses, to explore the feasibility of effective defocus micro lens design, and apply personalized defocus frame lenses for myopia prevention and control.

SUMMARY:
To evaluate the differences in controlling the progression of myopia in adolescents and the safety and comfort of wearing different types of defocus incorporated multiple segments spectacle lenses, to explore the feasibility of effective defocus micro lens design, and apply personalized defocus frame lenses for myopia prevention and control.

ELIGIBILITY:
Inclusion Criteria:

1. Age: 6-14 years old;
2. After using 1% cyclohexanone hydrochloride eye drops (Saifeijie) for ciliary muscle paralysis, binocular spherical power were within 0.00D~-4.00D, binocular cylinder power ≤ 1.50D, the anisometropia is less than 1.50D, and the best corrected visual acuity was above 5.0;
3. Within 30 days, the myopia prevention and control methods such as multifocal glasses, orthokeratology, defocusing flexible glasses, progressive glasses, atropine eye drops, red light and acupuncture and moxibustion treatment were not used;
4. The subject has a willingness to receive treatment and an informed consent form is signed by their legal guardian.

Exclusion Criteria:

1. Diagnosed constant strabismus;
2. Diagnosed pathological myopia;
3. Other congenital eye diseases;
4. Researchers believe that the patients have other reasons that are not suitable for inclusion in the project.

Ages: 6 Years to 14 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 252 (Estimated)
Dates: Start 2024-03-01 (Actual); Primary Completion 2025-06-30 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Axial length | 2 years
  The change of axial length.

SECONDARY OUTCOMES:
Subjective refraction equivalent spherical | 2 years
  The change of Subjective refraction equivalent spherical

CONTACTS AND LOCATIONS:
Locations (1):
- Shanghai Eye Diseases Prevention &Treatment Center/ Shanghai Eye Hospital, School of Medicine, Tongji University, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: No